CLINICAL TRIAL: NCT04407377
Title: A Randomized, 4-Period, Crossover Study to Investigate the Effects of Tolperisone on Measures of Drowsiness and Cognitive Function Compared to Cyclobenzaprine and Placebo
Brief Title: Effects of Tolperisone on Measures of Drowsiness and Cognitive Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurana Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLN-116
Record Dates: First submitted 2020-05-07; First posted 2020-05-29 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Healthy
MeSH Terms: interventions — Tolperisone; cyclobenzaprine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Tolperisone 200 mg (Experimental): Study Drug, Tolperisone 200mg TID
  Interventions: Drug: Tolperisone Hydrochloride
- Tolperisone 400 mg (Experimental): Study Drug, Tolperisone 400mg TID
  Interventions: Drug: Tolperisone Hydrochloride
- Cyclobenzaprine (Active Comparator): Active Comparator, Cyclobenzaprine 10mg TID
  Interventions: Drug: Cyclobenzaprine Hydrochloride 10 MG
- Placebo (Placebo Comparator): Placebo, TID
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tolperisone Hydrochloride — Study Drug
  Other Names: Tolperisone
  Arms: Tolperisone 200 mg; Tolperisone 400 mg
Drug: Cyclobenzaprine Hydrochloride 10 MG — Active Comparator
  Arms: Cyclobenzaprine
Other: Placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
A Randomized, 4-Period, Crossover Study to characterize the effects of tolperisone 200 mg and 400 mg (supratherapeutic dose) three times a day (TID) over 3 days of dosing on measures of simulated driving performance, cognitive function and drowsiness and compared to placebo and cyclobenzaprine (single-day, residual effect, multiple-day).

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory male or female, between 21 and 65 years of age, inclusive, for the entire duration of the study (from Screening through Day 3 of last treatment period).
* Body mass index (BMI) range between 18.5 and 30.0 kg/m2, inclusive.
* Subject must possess a valid driver's license and be an active driver and have driven a minimum of 10,000 miles (about 16,000 km) per year for the previous 3 years.
* Subject must demonstrate simulator sickness questionnaire scores that are not indicative of simulator sickness as defined in the driving simulation operations manual.
* Subject must have a regular sleep pattern, not be engaged in shift-work, and in general, have at least 7 hours of sleep each night.

Exclusion Criteria:

* History of sleep disorders, including insomnia, sleep apnea, Restless Legs Syndrome (RLS), or narcolepsy, night-shift workers, routine daytime napping or oversleeping on weekends days (off work) or a score higher than 10 on the Epworth Sleepiness Scale (ESS) at Screening.
* A history of difficulty in falling asleep or staying asleep in the previous 3 months that is considered clinically significant by the Investigator.
* Subject has traveled across 2 or more time zones (trans meridian travel) in the last 2 weeks prior to randomization or is expected to travel across 2 or more time zones during the study.
* Subject has any physical condition (e.g., severe vision issues, hand use limitations) that would prevent the subject from performing the cognitive or drowsiness assessments.
* Subject has a presence or history of any medically diagnosed, clinically significant psychiatric disorder, including depression, anxiety, insomnia, schizophrenia, or bipolar disorder.
* Consumes more than 3 cups of coffee per day.
* Female subjects who are pregnant or lactating.
* Any clinically significant medical abnormality, any clinically significant chronic disease, or any clinically significant finding on physical examination.
* Subject with a genotype status of poor-, ultrarapid-, or indeterminate- metabolizers of cytochrome CYP2D6.
* Subject is unable to remain in the research unit for each of the treatment periods.
* Subject has visual or auditory impairment which in the opinion of the Investigator would interfere with study related procedures or study conduct.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Driving Performance | Day 1
  Standard Deviation of Lateral Position, measured by simulated driving performance using Cognitive Research Corporation Driving Simulator-MiniSim (CRCDS-MiniSim), of tolperisone compared to placebo

SECONDARY OUTCOMES:
Karolinska Sleepiness Scale | Day 1
  Measure of Drowsiness
Epworth Sleepiness Scale | Day 3
  Measure of Drowsiness
Reaction Time | Day 1
  Measure of Cognitive Function
Rapid Visual Information Processing | Day 1
  Measure of Cognitive Function
CogScreen Symbol Digit Coding Test | Day 1
  Measure of Cognitive Function

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - CNS Trial, Long Beach, California
  - Hassman Research Institute, Berlin, New Jersey

IPD SHARING:
Plan to Share IPD: No